CLINICAL TRIAL: NCT05236023
Title: Evaluation of a Family-centred Care Intervention Based on Zero Separation and Couplet Care
Brief Title: Family Centred Healthcare - Zero Separation and Couplet Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Michella Runge Kjøbeløv Bjerregaard, Principal investigator, Copenhagen University Hospital, Hvidovre
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: P-2021-872
Record Dates: First submitted 2022-01-08; First posted 2022-02-11 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Premature Birth; Post Partum; Infant; Mother-Child Relations; Family
Keywords: preterm infants; zero-separation; Family centred care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Group receiving care as usual before the intervention takes place
- Intervention group (Experimental): Group receiving zero separation and couplet care
  Interventions: Behavioral: Zero separation and couplet care

INTERVENTIONS:
Behavioral: Zero separation and couplet care — The essence of the intervention is that treatment-requiring mother-infant dyads are admitted together and receives couplet care provided by neonatal nurses.
  The nurses will be educated for the intervention by participating in a two-day course about postpartum observations, treatment and care; and participate in education about family-centred care and family-focused nursing.
  Arms: Intervention group

SUMMARY:
Today mother and infant are routinely separated directly after birth if there is a need of specialised treatment and care, despite of the significant and positive effects of skin-to-skin contact. Thus, there is a need of change in organizing the treatment and care in a way that minimizes separation.

The aim is to evaluate the implementation and effect of a complex family-centred intervention based 107 on zero separation and couplet care.

The intervention is rooted in the philosophy of family-centred care. Essentially, mother infant dyads will be admitted together, where they will receive couplet care by neonatal nurses. The study comprises a quasi-experimental trial and a qualitative process evaluation including a field study and two interview studies. Finally, a health economic evaluation will be conducted to assess the cost-effectiveness of this complex intervention. The intervention will take place at the Neonatal Intensive Care Unit at Hvidovre Hospital. The nurses will as a part of the intervention be educated to take care of both mother and infant and carry out the intervention.

Five families with experiences from the Neonatal Intensive Care Unit and the Maternity Unit participates as patient and public representative in the project, as their experiences and ideas will provide an added value to the project.

This study contribute with a new perspective on how to organize the treatment and care of a newborn family in a Neonatal Intensive Care Unit. The study will be the first to examine zero separation and couplet care within sick mother-infant dyads. The study will provide knowledge about how an intervention consisting of zero separation and couplet care can be feasible and acceptable, and what kind of effect and impact it will provide. It is expected that the study as a whole may impact and profile clinical nursing, as well as benefitting public health.

DETAILED DESCRIPTION:
"There is no such thing as a baby, there is a baby and someone".

Approximately 10% of all newborn infants are admitted to a neonatal intensive care unit (NICU) for medical reasons and care, due to sickness related to birth or because of preterm delivery, defined as a live birth occurring before 37 weeks of gestation. In Denmark, around 60,000 infants are born per year. Having a sick or preterm infant is stressful and a considerable challenge for parents and in this context anxiety, depression and stress is often reported. Many mothers to infants born sick or premature have extended need of postpartum care and treatment and will because of this be separated from their newborn infant and admitted to the maternity unit (MU). Depending on the circumstances it can be hours or days before mother and infant are reunited. Mothers reports separation from their infant as one of the highest sources of stress. The first hours of an infant's life are of special importance, when the transition from the intra - to extra-uterine life takes place, as instability in this period may cause a cascade of negative effects. Early separation is found to have negative effects on interaction, child development and aggression level, respectively. The findings support the presence of a "early sensitive period" for both mother and infant. On the other hand, there is evidence of benefits from skin-to-skin contact immediately after birth as it improves growth and thermal control in the infant, breastfeeding initiation and duration, and the physiological bonding between mother and infant. The World Health Organization recommends infants and mothers, even with confirmed Covid19, to practice skin-to-skin contact as it supports health and wellbeing in the family. However, today mother and infant are still routinely separated directly after birth if there is need of specialised treatment and care, despite of the significant and positive effects of skin-to-skin contact. Thus, there is a need of a change in organizing the treatment and care of mother-infant dyads in a way that minimizes separation - with a goal of zero-separation. New healthcare models are necessary, and these should include the care of the family. Family centred care (FCC) has been a central philosophy of care for many years in paediatric healthcare and zero-separation can be obtained by FCC supplemented with a couplet care model, meaning that mother and infant are being treated as an inseparable unit, with care of both the sick postpartum mother and the sick infant in the same room, by the same nurse. Zero separation and couplet care has been successfully examined in Sweden and Canada, with positive reaction from parents, professionals, and the organization; however, they have primarily studied the concept in relatively well infants and mothers. Thus, there is a need of providing scientific knowledge on treatment and care for severe sick mother-infant dyads. Furthermore, there is a need of knowledge about how an intervention, consisting of the concepts of zero separation and couplet care can be feasible, acceptable, and sustainable, from the point of view of both families, professionals, and the healthcare organization. System changes, educational changes and substantial adjustment is needed, to ensure effective and safe care of both mother and infant.

Copenhagen University Hospital Amager Hvidovre (AHH) is the largest national delivery hospital in Denmark and has about 7,000 deliveries a year, approximately 12% of total annual Danish births. The NICU at AHH has around 1,000 admissions yearly with a wide range, from premature infants above gestational age 28 weeks and sick infants after birth. The mean admission in NICU are 7.1 days with a range from 24 hours to three months.The NICU will move into new facilities in 2023, with 23 family rooms where all mothers with mild to severe treatment-requiring conditions will be couplet care for by nurses, which will be innovative and unique compared to present national and international treatment and care models, where mother and infant is separated.

The aim is to evaluate the implementation and effect of a complex family-centred intervention based on zero separation and couplet care.

The study adheres to the framework of the Medical Research Council (MRC)20. We will comprehensively evaluate the intervention by combining a quasi-experimental trial for the effect evaluation and a qualitative process evaluation consisting of a field study and two interview studies. Finally, we will conduct a health economic evaluation.

The quasi-experimental trial investigates the effect of the intervention by comparing it with usual care with respect to:

1. Infant length of stay (LOS)
2. Infant first SSC with parents
3. Mother's first breast stimulation
4. Family health and wellbeing

The sample size is based on a clinically relevant reduction of LOS by one day for the intervention compared with the control group. In pre-existing LOS data collected in 2021 from the intervention setting, the distribution could not be assumed to be normal. Therefore, the sample size calculation is based on the Wilcoxon rank-sum test. Sample size is estimated by simulation based on 1,000 repetitions (mean: 10.7, median: 5, standard deviation: 12.5), using the pre-existing data as control and intervention data generated by shifting the control data down one day in LOS. This produced a sample size of 239 families in each group (P < 0.05; 80% power).

The qualitative process evaluation examines the context, implementation and mechanism of impact guided by MRC21, specifically:

1. Contextual factors and causal mechanisms
2. Fidelity, adoption, and reach
3. Acceptability and appropriateness

Finally, the health economic evaluation will assess:

a) The cost-effectiveness of implementing the intervention.

Ethics Participating families and healthcare professionals will be informed about the purpose of the project and will receive oral and written information about the project prior to participation. According to the Declaration of Helsinki data will be handled confidently and when publishing the participants will be anonymized and written informed content will be obtained from all participants. The project will be reported to 'Videnscenter for dataanmeldelser' through Pacticus. Data are collected in REDcap and personally identifiable data will be stored in a hospital servers logged drive. Further, the regional Committee on Health Research Ethics is contacted about the duty to notify the project to the committee.

Perspective This study contribute with a new perspective on how to organize the treatment and care of a newborn family in a Neonatal Intensive Care Unit. The study will be the first to examine zero separation and couplet care within sick mother-infant dyads. The study will provide knowledge about how an intervention consisting of zero separation and couplet care can be feasible and acceptable, and what kind of effect and impact it will provide. It is expected that the study as a whole may impact and profile clinical nursing, as well as benefitting public health.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with a treatment-requiring condition such as preeclampsia, bleeding, psychological diagnoses, discontinued milk production and infection.
* Infant from gestational age 28 weeks with a treatment-requiring condition such as respiratory distress syndrome (with respiratory support including mechanical ventilation), hyperbilirubinemia, infection, and low blood sugar.

Exclusion Criteria:

* Healthy mothers who does not need care and treatment, and has an infant admitted at NICU.
* Mothers who are admitted at an adult intensive care unit due to severe sickness (severe preeclampsia with spasm, severe bleeding of 4-5 liter, and severe HELLP syndrome) - counting one-two mothers a year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Lenght of stay | At discharge assessed up to 6 months
  Hours of admission from birth to discharge

SECONDARY OUTCOMES:
Skin-to-skin contact | Hours from birth to first skin-to-skin contact
  First skin-to-skin contact
First breast stimulation | within the first 3 days
  Number of hours until mothers first breast tension
Family centred care scale | At discharge assessed up to 6 months and four months after discharge
  Family Centered Nursing Scale consists of seven statements that focus on the way nurses work and whether the nurses' work is performed in accordance with the principles of Family Centered Nursing. 7 items using a 5 point scale from not at all important to very important.
Parental Stress Scale | At discharge assessed up to 6 months and four months after discharge
  Measures parental stress, 18 items, The item statements are rated for agreement by parents using a 5-point response scale (1 = strongly disagree, 2 = disagree, 3 = undecided, 4 = agree, 5 = strongly agree)
PedsQL family impact scale | At discharge assessed up to 6 months and four months after discharge
  PedsQL™ Family Impact Module was designed to measure the impact of pediatric chronic health conditions on parents and the family. The PedsQL™ Family Impact Module measures parent selfreported physical, emotional, social, and cognitive functioning, communication, and worry. 24 items, rates on a five point scale from never to almost.
The Edinburgh postnatal depression scale | At discharge assessed up to 6 months and four months after discharge
  The Edinburg Postnatal Depression Scale (EPDS) was developed to assess depressive symptoms in the perinatal period. It consists of ten items scored from zero to three with a maximum total score of 30. Higher scores indicate a higher risk of developing a depression

CONTACTS AND LOCATIONS:
Overall Officials: Anne Brødsgaard, Study Chair — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark